CLINICAL TRIAL: NCT04525105
Title: ARE SMAD2, SMAD3 AND TGF-β GENE EXPRESSION VALUABLE IN THE MANAGEMENT OF THE URGE URINARY INCONTINENCE?
Brief Title: SMAD2, SMAD3 AND TGF-β GENE EXPRESSION IN URGE URINARY INCONTINENCE
Status: Completed | Type: Observational
Sponsor: Muğla Sıtkı Koçman University (Other)
Responsible Party: Principal Investigator, Melike Nur AKIN, Dr Melike Nur Akın, Muğla Sıtkı Koçman University
Other Study IDs: 18/II/26.10.20
Record Dates: First submitted 2020-08-20; First posted 2020-08-25 (Actual); Last update posted 2020-08-25 (Actual); Status verified 2020-08

CONDITIONS: SMAD2; SMAD3; TGF-β; Pelvic Organ Prolapse; Urge Urinary Incontinence
MeSH Terms: conditions — Pelvic Organ Prolapse; Urinary Incontinence, Urge

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Study group: wıth URGE INCONTINANCE
  Interventions: Genetic: SMAD2
- Control group: not urge incontinance
  Interventions: Genetic: SMAD2

INTERVENTIONS:
Genetic: SMAD2 — a family of structurally related cytokines
  Other Names: SMAD3; TGF-β1

SUMMARY:
Urge urinary incontinence (UUI) is a common health problem. Changes in collagen metabolism in pelvic support organs, such as uterosacral ligaments (USLs), might be responsible for the complex pathophysiology of UUI. The TGF-β pathway is involved in collagen synthesis and degradation. The Transforming Growth Family- β (TGF-β) superfamily has essential intracellular signaling components, such as newly identified SMAD family members. We evaluated the changes in the levels of TGF-β and SMAD gene and protein expression in the USL of patients with concomitant pelvic organ prolapse (POP) and UUI.

DETAILED DESCRIPTION:
This study included 10 patients who had been diagnosed with POP and UUI in the study group and 14 asymptomatic women without complaints of POP and UUI in the control group. Biopsy samples were collected from bilateral USL tissues during vaginal or abdominal hysterectomy. Total RNA was extracted from USL tissue and analyzed by qPCR. The protein expression levels were also analyzed with ELISA.

ELIGIBILITY:
Inclusion Criteria:

* patients who had been diagnosed with POP and UUI
* asymptomatic women without complaints of POP and UUI

Exclusion Criteria:

* Women who have SUI,
* a history of gynecologic malignancy,
* endometriosis,
* connective tissue disorders,
* asthma,
* previous pelvic inflammatory disease,
* pelvic radiation anamnesis,
* smoking,
* previous surgery for POP or UI,
* those on steroid therapy and hormone replacement therapy

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — > 18 years
Study Population: patients who had been diagnosed with POP and UUI and asymptomatic women without complaints of POP and UUI
Sampling Method: Probability Sample
Enrollment: 24 (Actual)
Dates: Start 2017-11-01 (Actual); Primary Completion 2020-01-01 (Actual); Study Completion 2020-01-01 (Actual)

PRIMARY OUTCOMES:
SMAD2 | intraoperative
  tissue expression and protein level
SMAD3 | intraoperative
  tissue expression and protein level
TGF-ß1 mRNA Expression Levels | intraoperative
  tissue expression and protein level

CONTACTS AND LOCATIONS:
Locations (1):
- Mugla Sıtkı Kocman University Faculty of Medicine, Muğla, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Undecided
If anyone demand the results of our study, we can share data with other researchers

REFERENCES:
- [Derived] Akin MN, Sivaslioglu AA, Edgunlu T, Kasap B, Celik SK. SMAD2, SMAD3 and TGF-beta GENE expressions in women suffering from urge urinary incontinence and pelvic organ prolapse. Mol Biol Rep. 2021 Feb;48(2):1401-1407. doi: 10.1007/s11033-021-06220-4. Epub 2021 Feb 18. PMID 33599951